CLINICAL TRIAL: NCT06287047
Title: The Impact of Using Different Spinal Needle Sizes on the Efficacy of the Dural Puncture Epidural Block: Comparative Randomized Controlled Study
Brief Title: The Impact of Using Different Spinal Needle Sizes on the Efficacy of the Dural Puncture Epidural Block
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Reham Mahrous, Assistant professor, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Other
Other Study IDs: spinal needle sizes and DPE
Record Dates: First submitted 2024-02-23; First posted 2024-02-29 (Actual); Last update posted 2025-04-29 (Actual); Status verified 2025-04

CONDITIONS: Dural Puncture Epidural Technique
Keywords: Dura; Dural puncture; epidural
MeSH Terms: interventions — Analgesia, Epidural

STUDY DESIGN:
Intervention Model Description: 81 patients meeting the inclusion criteria will be randomly divided into three equal groups: Group A (n=27): Conventional epidural. Group B (n=27): Dural puncture epidural with 25-gauge spinal needle. Group C (n=27): Dural puncture epidural with 27-gauge spinal needle.
Who Masked: Participant, Investigator
Masking Description: The details of the series will be unknown to the investigators and the group assignment will be kept in asset of sealed envelopes each bearing only the case number on the outside. Prior to surgery the appropriate numbered envelope will be opened by the nurse, the card inside will determine the patient group.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Conventional epidural group (Active Comparator): Conventional epidural.
  .
  Interventions: Procedure: Epidural analgesia
- DPE-25G group (Active Comparator): Dural puncture epidural with 25-gauge spinal needle.
  Interventions: Procedure: Epidural analgesia
- DPE-27G group (Active Comparator): Dural puncture epidural with 27-gauge spinal needle.
  Interventions: Procedure: Epidural analgesia

INTERVENTIONS:
Procedure: Epidural analgesia — Epidural analgesia alone or with dural puncture with different sizes of spinal needles
  Other Names: Dural puncture

SUMMARY:
The aim of this study is to compare the dural puncture epidural technique (DPET) with either 25-gauge spinal needle or 27-gauge spinal needle versus conventional epidural technique and evaluate whether DPET improves onset and spread of labor analgesia and if there is a role of the usage of different sized needles as regards block efficiency and complications.

DETAILED DESCRIPTION:
* 81 patients primigravida parturients (ASA II) in active labor
* uncomplicated pregnancy
* Cephalic presentation
* Cervical dilatation <5 cm

Exclusion criteria:

* Allergy to local anesthetics.
* Bleeding disorders
* Low platelet count
* Local or systemic sepsis
* Prior surgery in lumbosacral spine
* Patient's refusal.

Eighty-one patients meeting the inclusion criteria were randomly divided into three equal groups:

Group CE (n=27): Conventional epidural. Group DPE-25 (n=27): Dural puncture epidural with 25-gauge spinal needle. Group DPE-27 (n=27): Dural puncture epidural with 27-gauge spinal needle.

Randomization was done by computer generated numbers and concealed by serially numbered, opaque and sealed envelopes. The details of the series were unknown to the investigators and the group assignment was kept in a set of sealed envelopes, each bearing only the case number on the outside.

Full medical and surgical history were taken. Laboratory investigations were revised. Visual analogue scale was educated to the patient before the start of the operation.

One liter of lactated Ringer's solution was infused IV over 15 min during the neuraxial procedure.

The procedure was performed in the seated position. Parturients with VAS < 5 were excluded.

The procedure was performed by a senior anesthesia resident.

Before administering medications through the epidural catheter, subarachnoid, intravascular and subdural placement had to be ruled out.

After 5 min of the first initial bolus dose, adequacy of analgesia was assessed.

Analgesia was considered adequate if VAS score is ≤3. Onset of analgesia was defined as from time of first bolus dose to time of achieving VAS ≤3.

Patient with VAS score >3; considered failed block and were excluded from the study.

Analgesia was evaluated by a blinded observer assessing visual analog scale (VAS) pain scores, onset of analgesia, sensory level, and motor blockade.

The primary outcome was the onset of analgesia (defined as duration from injection of the first initial epidural bolus to attainment of VAS <3).

Other data collected are:

1. Patients' demographic data.
2. Obstetrics data.
3. Onset of analgesia (attainment of VAS <3).
4. HR and MABP (baseline, every 5 minutes until 15 mins, a every 15 mins till 1 hour and then every 1 hour till delivery).
5. Visual analogue scale (VAS) with hemodynamics.
6. Assessment of sensory level after 30 mins of the block.
7. Assessment of Sacral block during the 1st 30 minutes.
8. Assessment of motor block through the modified bromage scale
9. Occurrence of side effects as: Hypotension, bradycardia, nausea, vomiting and pruritis ,PDPH, nerve injury.

ELIGIBILITY:
Inclusion Criteria:

* ASAI & II parturient in active labor
* Uncomplicated pregnancy with vertex presentation
* Willing to participate in the study.

Exclusion Criteria:

* Patient's refusal
* Coagulopathy (INR> 1.5 and platelets < 80,000)
* Allergy to local anesthetics.
* Prior surgery in lumbosacral spine.

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — Parturients
Enrollment: 81 (Actual)
Dates: Start 2021-01-01 (Actual); Primary Completion 2022-01-31 (Actual); Study Completion 2024-06-15 (Actual)

PRIMARY OUTCOMES:
Onset of analgesia | 20 minutes
  Duration from injection of the first initial epidural bolus dose to attainment of VAS <3

SECONDARY OUTCOMES:
Degree of analgesia | 5 hours
  Visual Analogue Score (0-10)

CONTACTS AND LOCATIONS:
Locations (1):
- Faculty of Medidcne, Cairo Univerisity, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: No